CLINICAL TRIAL: NCT06788860
Title: Efficacy of Ultrasound-Guided Tri-Directional Needle Knife Release for Trigger Finger
Brief Title: Efficacy of Ultrasound-Guided Needle Knife Release for Trigger Finger
Acronym: UG-NK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Maher Ismail Ahmed Elashmawy (Other)
Responsible Party: Sponsor-Investigator, Mohamed Maher Ismail Ahmed Elashmawy, Lecturer of Rheumatology, Physical Medicine and Rehabilitation, Mansoura University Hospital
Organization: Mansoura University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mansoura_UG-KN_TF
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Trigger Finger
Keywords: Trigger Finger; A1 Pulley Release; Ultrasound-Guided Technique
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Intervention Model Description: All participants will undergo ultrasound-guided tri-directional needle knife release for trigger finger treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ultrasound-Guided Tri-directional Needle Knife Release Group (Experimental): Participants will undergo ultrasound- guided tri-directional needle knife release for treatment of trigger finger. Local anesthesia using 3-5 ml of 1% lidocaine and 0.25% bupivacaine will be administered for patient comfort. This procedure involves precise ultrasound guidance to ensure accurate and safe dissection of the thickened A1-Pulley.
  Interventions: Procedure: Tri-directional Ultrasound-guided Needle Knife Release

INTERVENTIONS:
Procedure: Tri-directional Ultrasound-guided Needle Knife Release — This procedure involves ultrasound-guided tri-directional needle knife release for the treatment of trigger finger. Local anesthesia using 3-5 ml of 1% lidocaine and 0.25% bupivacaine will be administered for patient comfort. It aims to ensure precise tissue dissection while minimizing risks and improving outcomes.
  Device: Sonosite M-Turbo Ultrasound Machine with Linear Probe HFL38x (6-13 MHz) is used for real-time imaging during the procedure.

SUMMARY:
Efficacy of ultrasound-guided tri-directional needle knife release in treating patients with trigger finger. The study evaluates safety, effectiveness, and recovery outcomes of a minimally invasive procedure compared to conventional approaches.

DETAILED DESCRIPTION:
This is a clinical trial designed to investigate the efficacy and safety of ultrasound-guided tri-directional needle knife release in patients with trigger finger, especially those patients for whom conservative treatments have failed. Trigger finger is caused by of thickening of the A1 pulley, leading to pain and stiffness, which results in limitation of the hand. The procedure will be carried out under local anesthesia and guided by ultrasound to be very accurate and safe, avoiding all possible risks. Patients will be assessed for better improvement in hand functioning, pain scale basing on visual analog scale, and above all patient overall satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic TF at the level of A1 pulley
* Trigger finger of Green's grades II or III or IV (moderate to severe)
* Symptoms persist for at least three months despite conservative treatments.
* Ability to provide informed consent and comply with follow-up requirements.

Exclusion Criteria:

* Patients with secondary causes of TF like diabetes mellitus, rheumatoid arthritis, gout, hypothyroidism, amyloidosis, and sarcoidosis.
* Patients with TF of Green's grade I.
* Previous surgical intervention on the affected digit.
* Allergy or contraindication to local anesthetics.
* Pregnancy or lactation.
* Inability to comply with follow-up assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-10-29 (Estimated)

PRIMARY OUTCOMES:
Improvement in hand and finger function | 6 months
  Functional improvement evaluation using the QuickDASH score (0-100 scale)
Reduction in Pain scores post-procedure | 6 months
  Evaluating of the effectiveness of ultrasound-guided tri-directional needle knife release in reducing pain scores among patients with trigger finger using the Visual Analog Scale (VAS) (scale 0-10)
Improvement of finger mobility | 6 months
  Measurment of joint mobility in degrees at MCP and PIP joints using goniometer.

SECONDARY OUTCOMES:
Patient Satisfaction with the procedure | 6 months
  Evaluating of patient satisfaction levels using a structured questionnaire
Rate of procedure-related complications | 6 months
  Monitoring and documentation of procedure-related complications, including infection, nerve injury, and other adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant date (IPD) with other researchers.

REFERENCES:
- [Background] 1. Huisstede BM, Hoogvliet P, Coert JH, Fridén J, Group EH. Multidisciplinary consensus guideline for managing trigger finger: results from the European HANDGUIDE Study. Physical therapy. 2014;94(10):1421-33. 2. Ferrara PE, Codazza S, Maccauro G, Zirio G, Ferriero G, Ronconi G. Physical therapies for the conservative treatment of the trigger finger: a narrative review. Orthopedic Reviews. 2020;12(Suppl 1). 3. Lee SH, Choi YC, Kang HJ. Comparative study of ultrasonography-guided percutaneous A1 pulley release versus blinded percutaneous A1 pulley release. Journal of Orthopaedic Surgery. 2018;26(2):2309499018772368. 4. Sutter D, Treier A, Vögelin E. Sonographically controlled minimally-invasive A1 pulley release using a new guide instrument-a case series of 106 procedures in 64 patients. BMC musculoskeletal disorders. 2023;24(1):875. 5. Caballero EQ, Horcajadas ÁLB, Chaparro EC, Gana MDI, Franco IL-V, Villagrán JM. Ultrasound (US) of the fingers: anatomy and pathology. Quantitative Imaging in Medicine and Surgery. 2024;14(11):8012. 6. Pan M, Sheng S, Fan Z, Lu H, Yang H, Yan F, et al. Ultrasound-guided percutaneous release of A1 pulley by using a needle knife: a prospective study of 41 cases. Frontiers in Pharmacology. 2019;10:267. 7. Nikolaou VS, Malahias M-A, Kaseta M-K, Sourlas I, Babis GC. Comparative clinical study of ultrasound-guided A1 pulley release vs open surgical intervention in the treatment of trigger finger. World journal of orthopedics. 2017;8(2):163. 8. Langley G, Sheppeard H. The visual analogue scale: its use in pain measurement. Rheumatology international. 1985;5(4):145-8. 9. Kennedy CA, Beaton DE, Smith P, Van Eerd D, Tang K, Inrig T, et al. Measurement properties of the Quick DASH (disabilities of the arm, shoulder and hand) outcome measure and cross-cultural adaptations of the Quick DASH: A systematic review. Quality of life research. 2013;22:2509-47. 10. Wolfe SW. Tendinopathy. Green's operative hand surgery. 2011:2067-88.